CLINICAL TRIAL: NCT03028974
Title: Adaptive and Innate Immunity, Memory and Repertoire in Vaccination and Infection
Brief Title: Innate and Acquired Immunity to Influenza Infection and Immunization (SLVP029)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Cornelia L. Dekker, Professor, Pediatrics, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SU-31136-2014-2019; U19AI057229-11 (NIH)
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Results first posted 2018-12-14 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-11

CONDITIONS: Influenza
Keywords: Inactivated influenza vaccine; Live, attenuated influenza vaccine; Young children; Adults
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Group A: 2-4 yo LAIV4 (Return) (Other): Participants are given quadrivalent live, attenuated influenza vaccine (LAIV4)/ FluMist® . For children requiring 2 doses of vaccine, a second immunization will be given at Day 28-32 after Dose 1. All participants in this group will be asked to return annually for repeat immunization per ACIP guidelines and blood sample collection.
  Interventions: Biological: FluMist®
- Group B: 2-4 yo LAIV4 (Single Yr) (Other): Participants are given LAIV4/ FluMist® and participate for single year. For children requiring 2 doses of vaccine, a second immunization will be given at Day 28-32 after Dose 1.
  Interventions: Biological: FluMist®
- Group C: 2-4 yo LAIV4 (Swab/Single Yr) (Other): Participants are given LAIV4/ FluMist® and participate for single year. NP swabs are collected; no blood samples will be collected for this group. For children requiring 2 doses of vaccine, a second immunization will be given at least 28 days after Dose 1.
  Interventions: Biological: FluMist®
- Group D: 6 - 23 mos old IIV4 (Return) (Other): Participants are given a quadrivalent inactivated influenza vaccine (IIV4)/ Fluzone® . For children requiring 2 doses of vaccine (vaccine-naïve), a second immunization will be given at Day 28-32 after Dose 1. Participants are asked to return annually for repeat immunization per ACIP guidelines and blood sample collection.
  Interventions: Biological: Fluzone®
- Group E: 6 - 23 mos old IIV4 (Single Yr) (Other): Participants are given IIV4/ Fluzone® and participate for a single year. For children requiring 2 doses of vaccine (vaccine-naïve), a second immunization will be given at Day 28-32 after Dose 1.
  Interventions: Biological: Fluzone®
- Group F: 9-13/18-49 yo LAIV4 (Single Yr) (Other): Participants 9-13 year old and 18-49 year old are given LAIV4/ FluMist® . Participants will participate for a single year.
  Interventions: Biological: FluMist®
- Group G: 9-13/18-49 yo IIV4 (Single Yr) (Other): Participants 9-13 year old and 18-49 year old are given IIV4/ Fluzone® and participate for single year.
  Interventions: Biological: Fluzone®

INTERVENTIONS:
Biological: Fluzone® — Fluzone® Quadrivalent: Quadrivalent influenza virus vaccine
  Arms: Group D: 6 - 23 mos old IIV4 (Return); Group E: 6 - 23 mos old IIV4 (Single Yr); Group G: 9-13/18-49 yo IIV4 (Single Yr)
Biological: FluMist® — FluMist® Quadrivalent: Quadrivalent influenza virus vaccine live, intranasal spray
  Arms: Group A: 2-4 yo LAIV4 (Return); Group B: 2-4 yo LAIV4 (Single Yr); Group C: 2-4 yo LAIV4 (Swab/Single Yr); Group F: 9-13/18-49 yo LAIV4 (Single Yr)

SUMMARY:
The purpose of the study is to get a better understanding of the natural and adaptive immune response to the flu virus and to compare the immune cell responses to FDA-licensed flu vaccines in nasal mucosal cells and in blood.

DETAILED DESCRIPTION:
This is a study of healthy children and adults receive the current seasonal influenza vaccine. The volunteers were enrolled into one of 7 groups over a 5-year period. Immunization is administered; blood samples and NP swabs are collected at various time points based on groups assigned.

Group A (LAIV4/annual return): Up to six 2-4 year old volunteers are given a quadrivalent live, attenuated influenza vaccine (LAIV4). All participants in this group are asked to return annually for flu immunization and blood samples on Day 0 and Day 7 post immunization. Vaccine naive children returned 30 days later for a second immunization per standard of care. This group was discontinued in year 3 due to Advisory Committee on Immunization Practices (ACIP) recommendations against the use of LAIV.

Group B (LAIV4/ single year): Up to twenty 2-4 year old volunteers were given a quadrivalent live, attenuated influenza vaccine (LAIV4). Volunteers will participate for a single year. All participants in this group were immunized on Day 0. Blood samples were taken on on Day 0 and Day 7 post immunization. Vaccine naive children returned 30 days later for a second immunization per standard of care. This group was discontinued in year 3 due to ACIP recommendations against the use of LAIV.

Group C (LAIV4/NP swab group): Up to twenty 2-4 year old volunteers were given a quadrivalent live, attenuated influenza vaccine (LAIV4). Nasopharyngeal samples (NP) swabs were collected Day 1 and 21 and 28 post immunization. No blood was collected for this group. Vaccine naive children returned 30 days later for a second immunization per standard of care. This group was discontinued in year 3 due to ACIP recommendations against the use of LAIV.

Group D (IIV4/annual return): Up to six 6 month-23 month old (inclusive) volunteers are given a quadrivalent inactivated influenza vaccine (IIV4). All participants in this group are asked to return annually for flu immunization and blood samples on Day 0 and Day 7 post immunization. Vaccine naive children returned 30 days later for a second immunization per standard of care.

Group E (IIV4/single year): Up to twenty 6 month-23 month old (inclusive) volunteers were given a quadrivalent inactivated influenza vaccine (IIV4). Volunteers participate for a single year. All participants in this group were immunized on Day 0. Blood samples were taken on on Day 0 and Day 7 post immunization. Vaccine naive children returned 30 days later for a second immunization per standard of care.

Group F (LAIV4/single year) Up to forty 9-13 year old (n= 20) and 18-49 year old (n= 20) volunteers were given live, attenuated influenza vaccine (LAIV). Blood samples were collected Days 0, 7, and 28 and NP swabs were collected Days 1 and 28. This group was discontinued in year 3 due to ACIP recommendations against the use of LAIV.

Group G (IIV4/single year) Up to forty, 9-13 year old (n= 20) and 18-49 year old (n= 20) volunteers were given a quadrivalent inactivated influenza vaccine (IIV4). Blood samples were collected Day 0,7, and 28

ELIGIBILITY:
Inclusion Criteria:

1. Otherwise healthy, 6 mo-49 year-old volunteers.
2. Willing to complete the informed consent process (including assent for minors 7-17 years of age).
3. Availability for follow-up for the planned duration of the study.
4. For parents of children 6 months - 4 years of age: Willing to participate in the study annually for up to 5 years (if yes, consider for annual return groups).
5. Acceptable medical history by review of inclusion/exclusion criteria and vital signs.
6. Influenza vaccine-naive or only one prior season of flu immunization with IIV (does not apply to Groups F and G).

Exclusion Criteria:

1. Prior off-study vaccination with the current year's seasonal influenza vaccine
2. Receipt of LAIV in the prior season (does not apply to Groups F and G)
3. Received flu immunizations in 2 or more prior flu seasons (does not apply to Groups F and G)
4. Allergy to egg or egg products, or to vaccine components, (including gentamicin, gelatin, arginine or MSG if given LAIV4)
5. Life-threatening reactions to previous influenza vaccinations
6. Asthma in adults. Children aged 2 through 4 years who have asthma or who have had a wheezing episode noted in the medical record within the past 12 months, or for whom parents report that a health care provider stated that they had wheezing or asthma within the last 12 months [If yes, not eligible for LAIV Groups A, B, C, & F].
7. Active systemic or serious concurrent illness, including febrile illness on the day of vaccination
8. History of immunodeficiency (including HIV infection)
9. For children or adolescents through 17 years of age,receiving aspirin therapy or aspirin-containing products [If yes, not eligible for LAIV Groups A, B, C, and F].
10. Known or suspected impairment of immunologic function, including, but not limited to, clinically significant liver disease, diabetes mellitus treated with insulin, moderate to severe renal disease, or any other chronic disorder which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
11. Blood pressure >150 systolic or >95 diastolic at first study visit and the day of vaccination (for children 12 yrs and older, and adults).
12. Hospitalization in the past year for congestive heart failure or emphysema.
13. Chronic Hepatitis B or C
14. Recent or current use of immunosuppressive medication, including systemic glucocorticoids (corticosteroid nasal sprays and topical steroids are permissible in all groups; inhaled steroid use is not permissible)
15. Participants in close contact with anyone who has a severely weakened immune system and requires a protective environment. Exposure to such persons should be avoided for 7 days after receipt of LAIV. [If yes, may be ineligible for Groups A,B, C and F].
16. Malignancy, other than squamous cell or basal cell skin cancer (includes solid tumors such as breast cancer or prostate cancer with recurrence in the past year, and any hematologic cancer such as leukemia).
17. Autoimmune disease (including rheumatoid arthritis treated with immunosuppressive medication such as Plaquenil, methotrexate, prednisone, Enbrel) which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol
18. History of blood dyscrasias, renal disease, or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year
19. Use of any anti-coagulation medication such as Coumadin or Lovenox, or anti-platelet agents such as aspirin (except up to 325 mg. per day), Plavix, or Aggrenox must be reviewed by investigator to determine if this would affect the volunteer's safety.
20. Has taken an influenza antiviral medication within 48 hours prior to study vaccination [If yes, not eligible for LAIV Groups A, B, C and F].
21. Receipt of blood or blood products within the past 6 months or planned used during the study
22. Medical or psychiatric condition or occupational responsibilities that preclude participant compliance with the protocol.
23. Receipt of inactivated vaccine 14 days prior to study enrollment, or planned vaccinations prior to completion of last study visit
24. Receipt of live, attenuated vaccine within 60 days prior to enrollment of planned vaccination prior to completion of last study visit
25. Need for allergy immunization (that cannot be postponed) during the study period
26. History of Guillain-Barre syndrome
27. Pregnant woman
28. Breastfeeding [If yes, not eligible for LAIV Group F]
29. Use of investigational agents within 30 days prior to enrollment or planned use during the study
30. Donation of the equivalent of a unit of blood within 6 weeks prior to enrollment or planned donation prior to completion of the last visit
31. Any condition which, in the opinion of the investigator, might interfere with volunteer safety, study objectives or the ability of the participant to understand or comply with the study protocol.

Ages: 6 Months to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 77 (Actual)
Dates: Start 2014-09-17 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Dekker, MD, Principal Investigator — Stanford University; Harry Greenberg, MD, Principal Investigator — Stanford University; Xiaosong He, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants are presented only in the group in the year in which they received the vaccination. Planned Groups B and C did not enroll in years 2014-2018, Group A did not enroll in 2015-2018 and Group F did not enroll in years 2016-2018 due to LAIV not being recommended.
Groups:
- Group B: 2-4 yo LAIV4 (Single Year): Participants are given LAIV4/ FluMist® and participate for single year. For children requiring 2 doses of vaccine, a second immunization will be given at Day 28-32 after Dose 1.
  FluMist®: FluMist® Quadrivalent: Quadrivalent influenza virus vaccine live, intranasal spray
- Group D: 6 - 23 Mos Old IIV4 (Returning): Participants are given a quadrivalent inactivated influenza vaccine (IIV4)/ Fluzone® . For children requiring 2 doses of vaccine (vaccine-naïve), a second immunization will be given at Day 28-32 after Dose 1. Participants are asked to return annually for repeat immunization per ACIP guidelines and blood sample collection.
  Fluzone®: Fluzone® Quadrivalent: Quadrivalent influenza virus vaccine
Period: 2014-2015
Arm/Group | Group A: 2-4 yo LAIV4 (Return) | Group B: 2-4 yo LAIV4 (Single Year) | Group C: 2-4 yo LAIV4 (Swab/Single Yr) | Group D: 6 - 23 Mos Old IIV4 (Returning) | Group E: 6 - 23 Mos Old IIV4 (Single Yr) | Group F: 9-13/18-49 yo LAIV4 (Single Yr) | Group G: 9-13/18-49 yo IIV4 (Single Yr)
Started (LAIV was not recommended in Group B and C age groups starting in 2014-2015.) | 1 | 0 | 0 | 3 | 0 | 11 | 13
Completed | 1 | 0 | 0 | 3 | 0 | 11 (2 participants did not continue to the next period.) | 13 (13 participants did not continue to the next period.)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: 2015-2016
Arm/Group | Group A: 2-4 yo LAIV4 (Return) | Group B: 2-4 yo LAIV4 (Single Year) | Group C: 2-4 yo LAIV4 (Swab/Single Yr) | Group D: 6 - 23 Mos Old IIV4 (Returning) | Group E: 6 - 23 Mos Old IIV4 (Single Yr) | Group F: 9-13/18-49 yo LAIV4 (Single Yr) | Group G: 9-13/18-49 yo IIV4 (Single Yr)
Started (LAIV was not recommended in Groups A, B, C and F in 2015-2016.) | 0 | 0 | 0 | 6 (One participant joined from Group A, 2 new were enrolled.) | 0 | 14 (10 new participants were enrolled; 4 subjects switched from Group G.) | 20 (11 new participants were enrolled; 9 subjects switched from Group F.)
Completed | 0 | 0 | 0 | 6 (3 participants did not continue to the next period. 1 Participant returned in period 4 (2017-2018).) | 0 | 14 (14 participants did not continue to the next period.) | 20 (20 participants did not continue to the next period.)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: 2016-2017
Arm/Group | Group A: 2-4 yo LAIV4 (Return) | Group B: 2-4 yo LAIV4 (Single Year) | Group C: 2-4 yo LAIV4 (Swab/Single Yr) | Group D: 6 - 23 Mos Old IIV4 (Returning) | Group E: 6 - 23 Mos Old IIV4 (Single Yr) | Group F: 9-13/18-49 yo LAIV4 (Single Yr) | Group G: 9-13/18-49 yo IIV4 (Single Yr)
Started (Groups A, B, C and F closed to enrollment. LAIV4 not recommended.) | 0 | 0 | 0 | 4 (1 new participant was enrolled.) | 2 (2 new participants were enrolled.) | 0 | 18 (18 new participants were enrolled.)
Completed | 0 | 0 | 0 | 4 | 2 (2 participants did not continue to the next period) | 0 | 18 (18 participants did not continue to the next period.)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: 2017-2018
Arm/Group | Group A: 2-4 yo LAIV4 (Return) | Group B: 2-4 yo LAIV4 (Single Year) | Group C: 2-4 yo LAIV4 (Swab/Single Yr) | Group D: 6 - 23 Mos Old IIV4 (Returning) | Group E: 6 - 23 Mos Old IIV4 (Single Yr) | Group F: 9-13/18-49 yo LAIV4 (Single Yr) | Group G: 9-13/18-49 yo IIV4 (Single Yr)
Started | 0 | 0 | 0 | 5 | 0 | 0 | 5 (5 new participants were enrolled.)
Completed | 0 | 0 | 0 | 5 | 0 | 0 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: In 2014, LAIV was not recommended in this age group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: 2-4 yo LAIV4 (Return) | Group D: 6 - 23 Mos Old IIV4 (Return) | Group E: 6 - 23 Mos Old IIV4 (Single Yr) | Group F: 9-13/18-49 yo LAIV4 (Single Yr) | Group G: 9-13/18-49 yo IIV4 (Single Yr) | Total
Number analyzed (Participants) | 1 | 6 | 2 | 21 | 47 | 77
Age, Continuous [Median (Standard Deviation); unit: years] | 2 (0) | 1.5 (00.187) | 1 (0) | 20 (13.05) | 33.5 (1.48) | 21.1 (1.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 0 | 11 | 30 | 44
  Male | 1 | 3 | 2 | 10 | 17 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 1 | 6 | 2 | 19 | 45 | 73
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 6 | 12 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1 | 2
  White | 0 | 6 | 0 | 10 | 26 | 42
  More than one race | 1 | 0 | 0 | 3 | 8 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 6 | 2 | 21 | 47 | 77

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants From Each Arm Who Received Influenza Vaccine
Time Frame: Day 0 to 28-32 post immunization
Population: Participants with available data at the respective timepoint are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: 2-4 yo LAIV4 (Return) | Group D: 6 - 23 Mos Old IIV4 (Returning) | Group E: 6 - 23 Mos Old IIV4 (Single Yr) | Group F: 9-13/18-49 yo LAIV4 (Single Yr) | Group G: 9-13/18-49 yo IIV4 (Single Yr)
Number analyzed (Participants) | 1 | 7 | 2 | 25 | 56
Participants
  2014-2015: number analyzed (Participants) | 1 | 3 | 0 | 11 | 13
  2014-2015 | 1 | 3 |  | 11 | 13
  2015-2016: number analyzed (Participants) | 0 | 6 | 0 | 14 | 20
  2015-2016 |  | 6 |  | 14 | 20
  2016-2017: number analyzed (Participants) | 0 | 4 | 2 | 0 | 18
  2016-2017 |  | 4 | 2 |  | 18
  2017-2018: number analyzed (Participants) | 0 | 5 | 0 | 0 | 5
  2017-2018 |  | 5 |  |  | 5

2. Secondary Outcome: Count of Participants With Related Adverse Events
Time Frame: Day 0 to 28-32 post-immunization
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: 2-4 yo LAIV4 (Return) | Group D: 6 - 23 Mos Old IIV4 (Return) | Group E: 6 - 23 Mos Old IIV4 (Single Yr) | Group F: 9-13/18-49 yo LAIV4 (Single Yr) | Group G: 9-13/18-49 yo IIV4 (Single Yr)
Number analyzed (Participants) | 1 | 7 | 2 | 25 | 56
Participants | 0 | 1 | 0 | 7 | 4

ADVERSE EVENTS:
Time Frame: Day 0 to 28-32 post-immunization
Description: Only related adverse events and related serious adverse events were collected.
Groups:
- Group A: 2-4 yo LAIV4 (Return): Participants were given quadrivalent live, attenuated influenza vaccine (LAIV4)/ FluMist® . For children requiring 2 doses of vaccine, a second immunization was given at Day 28-32 after Dose 1. All participants in this group was asked to return annually for repeat immunization per ACIP guidelines and blood sample collection.
  FluMist®: FluMist® Quadrivalent: Quadrivalent influenza virus vaccine live, intranasal spray
- Group D: 6 - 23 Mos Old IIV4 (Returning): Participants were given a quadrivalent inactivated influenza vaccine (IIV4)/ Fluzone® . For children requiring 2 doses of vaccine (vaccine-naïve), a second immunization was given at Day 28-32 after Dose 1. Participants were asked to return annually for repeat immunization per ACIP guidelines and blood sample collection.
  Fluzone®: Fluzone® Quadrivalent: Quadrivalent influenza virus vaccine
- Group E: 6 - 23 Mos Old IIV4 (Single Yr): Participants were given IIV4/ Fluzone® and participate for a single year. For children requiring 2 doses of vaccine (vaccine-naïve), a second immunization was given at Day 28-32 after Dose 1.
  Fluzone®: Fluzone® Quadrivalent: Quadrivalent influenza virus vaccine
- Group F: 9-13/18-49 yo LAIV4 (Single Yr): Participants 9-13-year-old and 18-49-year-old were given LAIV4/ FluMist ®. Participants participated for a single year.
  FluMist®: FluMist® Quadrivalent: Quadrivalent influenza virus vaccine live, intranasal spray
- Group G: 9-13/18-49 yo IIV4 (Single Yr): Participants 9-13-year-old and 18-49-year-old were given IIV4/ Fluzone® and participated for a single year.
  Fluzone®: Fluzone® Quadrivalent: Quadrivalent influenza virus vaccine
Arm/Group | Group A: 2-4 yo LAIV4 (Return) | Group D: 6 - 23 Mos Old IIV4 (Returning) | Group E: 6 - 23 Mos Old IIV4 (Single Yr) | Group F: 9-13/18-49 yo LAIV4 (Single Yr) | Group G: 9-13/18-49 yo IIV4 (Single Yr)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/7 | 0/2 | 0/25 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/7 | 0/2 | 0/25 | 0/56
Other Adverse Events (participants affected / at risk) | 0/1 | 1/7 | 0/2 | 7/25 | 4/56
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: 2-4 yo LAIV4 (Return) (N=1) | Group D: 6 - 23 Mos Old IIV4 (Returning) (N=7) | Group E: 6 - 23 Mos Old IIV4 (Single Yr) (N=2) | Group F: 9-13/18-49 yo LAIV4 (Single Yr) (N=25) | Group G: 9-13/18-49 yo IIV4 (Single Yr) (N=56)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Mild Headache (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Rash with erythema below injection site
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ecchymosis (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Ecchymosis at phlebotomy site
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Post procedure bleeding (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — A small amount of blood noted on the swab when the NP sample was obtained.
Nasal mucous drainage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The original design of this study was corrupted when the ACIP decided that LAIV administration was not recommended over concerns re: decreased immunogenicity and effectiveness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT03028974/Prot_SAP_000.pdf